CLINICAL TRIAL: NCT06194864
Title: A Phase 1, Sequential Drug Interaction Study to Evaluate the Effect of CYP3A4 and P-glycoprotein Inhibition by Itraconazole or Induction by Rifampicin on the Pharmacokinetics of Ecopipam and Its Metabolites in Healthy Subjects
Brief Title: Drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emalex Biosciences Inc. (Industry)
Collaborators: Syneos Health (Other); Cambridge Cognition Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EBS-101-HV-106
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Drug Interaction
MeSH Terms: interventions — Itraconazole; Rifampin; ecopipam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): ecopipam 89.6 mg on Days 1 and 9 with repeat doses of itraconazole Days 6-16.
  Interventions: Drug: Itraconazole; Drug: Ecopipam
- Part 2 (Experimental): ecopipam 179.2 mg on Days 1 and 13 with repeat doses of rifampicin days 6-20.
  Interventions: Drug: rifampicin; Drug: Ecopipam

INTERVENTIONS:
Drug: Itraconazole — itraconazole 200 mg QD Days 6 to 16
  Arms: Part 1
Drug: rifampicin — rifampicin 600 mg QD Days 6 to 20
  Arms: Part 2
Drug: Ecopipam — 89.6 mg on Days 1 and 9 for Part 1 or 179.2 mg on Days 1 and 13 for Part 2

SUMMARY:
This is a single center, 2-Part, Phase 1, open-label, fixed-sequence, drug-drug interaction study designed to compare the PK of ecopipam when administered alone and in combination with itraconazole (Part 1) or rifampicin (Part 2) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects or femail subjects of non-childbearing potential
* ≥18 and ≤55 years of age
* BMI >18.5 and <30.0 kg/m2 and body weight ≥50.0 kg for males and ≥45.0 kg for females.
* Subjects must be healthy, as determined by the Investigator, based on medical history, physical examination, ECG, vital signs, and standard panel of blood and laboratory tests at Screening.
* Sexually active males must use a double barrier method of contraception during the study and for at least 90 days after the last dose of study drug.
* Male subjects must be willing not to donate sperm until 90 days following the last study drug administration.
* Willing to take off dentures or mouth piercing at the time of dosing.

Exclusion Criteria:

* History of significant medical illness
* Clinically significant abnormalities on screening tests/exams
* History of or significant risk of committing suicide
* Donation of plasma within 7 days prior to dosing
* Donation or significant loss of blood within 8 weeks prior to the first dosing
* Major surgery within 3 months or minor surgery within 1 month prior to admission
* Use of prohibited prescription, over-the-counter medications or natural health products
* Female subjects who are currently pregnant or lactating
* Positive pregnancy test
* Positive urine drug screen, urine cotinine test, or alcohol breath test
* Use of tobacco or nicotine products within 1 month prior to Screening
* Significant alcohol consumption
* History of drug abuse within the previous year, or a positive drug screen
* History of allergy to study medications
* Part 1 only: Presence of orthodontic braces or orthodontic retention wires
* Recent participation in a clinical research study
* Not suitable for study in the opinion of the Principal Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
AUC0-inf of ecopipam when administered with itraconazole | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-inf of ecopipam when administered without itraconazole | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-inf of ecopipam when administered with rifampicin | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-inf of ecopipam when administered without rifampicin | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-t of ecopipam when administered with itraconazole | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-t of ecopipam when administered without itraconazole | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-t of ecopipam when administered with rifampicin | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-t of ecopipam when administered without rifampicin | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of ecopipam when administered with itraconazole | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of ecopipam when administered without itraconazole | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of ecopipam when administered with rifampicin | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of ecopipam when administered without rifampicin | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
T½ el of ecopipam when administered with itraconazole | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
T½ el of ecopipam when administered without itraconazole | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
T½ el of ecopipam when administered with rifampicin | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
T½ el of ecopipam when administered without rifampicin | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis

SECONDARY OUTCOMES:
AUC0-inf of EBS-101-40853 | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-inf of ecopipam glucuronide | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-inf of EBS-101-40853 glucuronide | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-t of EBS-101-40853 | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-t of ecopipam glucuronide | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-t of EBS-101-40853 glucuronide | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of EBS-101-40853 | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of ecopipam glucuronide | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
Cmax of EBS-101-40853 glucuronide | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
T½ el of EBS-101-40853 | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
T½ el of ecopipam glucuronide | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
T½ el of EBS-101-40853 glucuronide | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-4 for ecopipam | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-4 for EBS-101-40853 | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-4 for ecopipam glucuronide | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
AUC0-4 for EBS 101-40853 glucuronide | Up to Day 21
  Up to 38 samples will be collected at the indicated time points for pharmacokinetic analysis
Minimum Modified Observer's Assessment of Alertness/Sedation (MOAA/S) score | Up to Day 21
  Score from 0-5 where 0 is no response and 5 is responds readily. MOAA/S measures will be recorded at the indicated timepoints
AUEC for Visual Analogue Scale (VAS) | Up to Day 21
  Score from 0 - 100 where 0 is not sedated and 100 is very sedated. VAS measures will be recorded at the indicated timepoints.
Maximum sedation for Visual Analogue Scale (VAS) | Up to Day 21
  Score from 0 - 100 where 0 is not sedated and 100 is very sedated. VAS measures will be recorded at the indicated timepoints.
AUEC for Reaction Time Index (RTI) score | Up to Day 21
  Reaction time for subject to release the response button after presentation of target stimulus.
Maximum sedation for Reaction Time Index (RTI) score | Up to Day 21
  Reaction time for subject to release the response button after presentation of target stimulus.
Safety and tolerability as demonstrated by AEs with itraconazole | Up to Day 30
  Subjects will be continually monitored for adverse events
Safety and tolerability as demonstrated by AEs without itraconazole | Up to Day 30
  Subjects will be continually monitored for adverse events
Safety and tolerability as demonstrated by AEs with rifampicin | Up to Day 30
  Subjects will be continually monitored for adverse events
Safety and tolerability as demonstrated by AEs without rifampicin | Up to Day 30
  Subjects will be continually monitored for adverse events
Safety and tolerability as demonstrated by Systolic blood pressure (SBP) and diastolic blood pressure (DBP) with itraconazole (mmHG) | Up to Day 21
  Blood pressure will be assessed as part of vital signs
Safety and tolerability as demonstrated by Systolic blood pressure (SBP) and diastolic blood pressure (DBP) without itraconazole(mmHG) | Up to Day 21
  Blood pressure will be assessed as part of vital signs
Safety and tolerability as demonstrated by Systolic blood pressure (SBP) and diastolic blood pressure (DBP) with rifampicin(mmHG) | Up to Day 21
  Blood pressure will be assessed as part of vital signs
Safety and tolerability as demonstrated by Systolic blood pressure (SBP) and diastolic blood pressure (DBP) without rifampicin(mmHG) | Up to Day 21
  Blood pressure will be assessed as part of vital signs
Heart rate with itraconazole (beats/minute) | Up to Day 21
  Heart rate will be assessed as part of vital signs
Heart rate without itraconazole (beats/minute) | Up to Day 21
  Heart rate will be assessed as part of vital signs
Heart rate with rifampicin (beats/minute) | Up to Day 21
  Heart rate will be assessed as part of vital signs
Heart rate without rifampicin (beats/minute) | Up to Day 21
  Heart rate will be assessed as part of vital signs
Respiratory rate pressure with itraconazole (breaths/minute) | Up to Day 21
  Respiratory rate will be assessed as part of vital signs
Respiratory rate without itraconazole (breaths/minute) | Up to Day 21
  Respiratory rate will be assessed as part of vital signs
Respiratory rate with rifampicin (breaths/minute) | Up to Day 21
  Respiratory rate will be assessed as part of vital signs
Respiratory rate without rifampicin (breaths/minute) | Up to Day 21
  Respiratory rate will be assessed as part of vital signs
Oral temperature with itraconazole (degrees Celsius) | Up to Day 21
  Temperature will be assessed as part of vital signs
Oral temperature without itraconazole (degrees Celsius) | Up to Day 21
  Temperature will be assessed as part of vital signs
Oral temperature with rifampicin (degrees Celsius) | Up to Day 21
  Temperature will be assessed as part of vital signs
Oral temperature without rifampicin (degrees Celsius) | Up to Day 21
  Temperature will be assessed as part of vital signs
Electrocardiogram (ECG) parameters: PR, RR, QRS, QT, and QT interval corrected for heart rate using Fridericia's formula (QTcF) with itraconazole (Milliseconds) | Up to Day 21
  Twelve-lead ECGs will be obtained at the indicated timepoints
Electrocardiogram (ECG) parameters: PR, RR, QRS, QT, and QT interval corrected for heart rate using Fridericia's formula (QTcF) without itraconazole (Milliseconds) | Up to Day 21
  Twelve-lead ECGs will be obtained at the indicated timepoints
Electrocardiogram (ECG) parameters: PR, RR, QRS, QT, and QT interval corrected for heart rate using Fridericia's formula (QTcF) with rifampicin (Milliseconds) | Up to Day 21
  Twelve-lead ECGs will be obtained at the indicated timepoints
Electrocardiogram (ECG) parameters: PR, RR, QRS, QT, and QT interval corrected for heart rate using Fridericia's formula (QTcF) without rifampicin (Milliseconds) | Up to Day 21
  Twelve-lead ECGs will be obtained at the indicated timepoints
Safety and tolerability as demonstrated by the Columbia Suicide Severity Rating Scale (C-SSRS) | Up to Day 21
  C-SSRS to be administered at the indicated timepoints
Values of white blood cell (WBC), neutrophils, lymphocytes, monocytes, eosinophils, basophils and platelets (1000/mm3) | Up to Day 21
  Blood samples will be collected for the assessment of hematology parameters
Value of hematocrit (percent) | Up to Day 21
  Blood samples will be collected for the assessment of hematology parameters
Value of hemoglobin (g/dL) | Up to Day 21
  Blood samples will be collected for the assessment of hematology parameters
Red blood cell (RBC) count (M/mm3) | Up to Day 21
  Blood samples will be collected for the assessment of hematology parameters
Values of sodium, potassium, chloride (mmol/L) | Up to Day 21
  Blood samples will be collected for the assessment of clinical chemistry parameters
Values of urea, phosphorus, calcium, glucose, and total, direct and indirect bilirubin (mg/dL) | Up to Day 21
  Blood samples will be collected for the assessment of clinical chemistry parameters
Values of albumin and total protein (g/dL) | Up to Day 21
  Blood samples will be collected for the assessment of clinical chemistry parameters
Values of alanine aminotransferase (ALT), aspartate aminotransferase (AST),alkaline phosphatase (ALP), gamma glutamyl transferase (GGT), creatininephosphokinase (CPK), and creatinine (U/L) | Up to Day 21
  Blood samples will be collected for the assessment of clinical chemistry parameters
Values of urine specific gravity | Up to Day 21
  Urine samples will be collected for the assessment of urine parameters
Values of urine pH | Up to Day 21
  Urine samples will be collected for the assessment of urine parameters
Values of urine glucose | Up to Day 21
  Urine samples will be collected for the assessment of urine parameters
Values of urine protein | Up to Day 21
  Urine samples will be collected for the assessment of urine parameters
Values of urine blood | Up to Day 21
  Urine samples will be collected for the assessment of urine parameters
Values of urine ketones | Up to Day 21
  Urine samples will be collected for the assessment of urine parameters
Values of urine bilirubin and nitrite | Up to Day 21
  Urine samples will be collected for the assessment of urine parameters
Values of urobilinogen | Up to Day 21
  Urine samples will be collected for the assessment of urine parameters
Values of urine leukocyte esterase by dipstick | Up to Day 21
  Urine samples will be collected for the assessment of urine parameters

CONTACTS AND LOCATIONS:
Overall Officials: Rick Munschauer, MSc, MD, FAAN, Study Director — Emalex Biosciences
Locations (1):
- Syneos Health Clinic Inc., Québec, Quebec, Canada